CLINICAL TRIAL: NCT03716544
Title: Efficacy of Amplification With Hearing Aids for Tinnitus Relief: a Randomized Controlled Trial
Brief Title: Efficacy of Amplification With Hearing Aids for Tinnitus Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, KAM Chi Shan Anna, Associate Professor, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RGC18100117
Record Dates: First submitted 2018-10-17; First posted 2018-10-23 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Tinnitus, Subjective; Hearing Impairment
Keywords: Tinnitus; Hearing Loss; Amplification; Sound Therapy
MeSH Terms: conditions — Tinnitus; Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Waiting list control group (No Intervention): There will be no treatment for 12 months.
- Hearing aid group (Experimental): Participants will receive amplification with hearing aids. Bilateral open-fit hearing aids will be fitted. Participants will be required to use the hearing aids for at least 2 hours daily for 12 months.
  Interventions: Device: Amplification with hearing aid
- Customized music group (Active Comparator): Customized music according to participants hearing level will be made available in an iPod. The iPod will deliver ear-specific therapeutic sound for asymmetrical hearing profile. Participants will have to listen to the therapeutic sound at a comfortable volume for two hours daily for 12 months.
  Interventions: Device: Customized music

INTERVENTIONS:
Device: Amplification with hearing aid — Use of hearing aids
  Other Names: Hearing aid group
  Arms: Hearing aid group
Device: Customized music — Customized music delivered via an iPod
  Arms: Customized music group

SUMMARY:
This study evaluates the treatment efficacy of tinnitus in people with mild hearing loss. One-third of participants will use hearing aid, one-third of participants will use customized music, while the other one-third participants will receive no treatment (waiting list control).

DETAILED DESCRIPTION:
Acoustic stimulation could induce plastic changes in the auditory cortex, and tinnitus mechanisms have been viewed as a negative consequence of neural plasticity in the central nervous system after peripheral aggression. Cortical changes (neural activity in the deafferented cortical area was reduced but the adjacent frequencies of the hearing loss region activated more extensive cortical areas) occur after sensorineural hearing loss, while exposure to an acoustically enriched environment or using hearing aids may minimize or reverse the plastic tonotopic map changes in the auditory cortex. The use of hearing aids in tinnitus management for people with significant hearing loss will always be associated with an improvement in hearing handicap and quality of life, and that complicates the interpretation of how much hearing aids specifically affect tinnitus. Thus studies on tinnitus patients with mild hearing loss could be illuminating, and this population will be targeted in the present study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or above
* can provide written informed consent
* have a diagnosis of subjective tinnitus, i.e., the tinnitus can only be heard by the patient and there is no acoustic source
* a tinnitus duration of more than one year
* have pure-tone average between 20 and 40 dB HL
* have bilateral symmetrical hearing loss (i.e. difference less than 15 dB)
* have at least a medium level of distress caused by tinnitus as indicated with total scores above 30 on the TQ-CH
* are committed to complete the 12-month follow-up

Exclusion Criteria:

* objective tinnitus, i.e. tinnitus produced by an internal acoustic source activating the cochlea and can be heard by another person
* received other forms of tinnitus treatments within three months before the baseline assessment session
* any history suggestive of psychiatric illness
* psychological distress or depression as indicated with total scores at or above 15 on the Cantonese HADS
* current hearing aid users
* inability to complete the study as revealed by the medical reports

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The Tinnitus Functional Index (Chinese version) (TFI-CH) | Change from baseline value at 3 months, 6 months and 12 months after the first day of treatment will be measured.
  TFI-CH is a 25-item self-administered questionnaire which assesses eight domains of tinnitus impact: intrusiveness; sense of control; cognitive; sleep; auditory; relaxation; quality of life (QoL); emotion. The total TFI score ranges 0 - 100, the higher score is indicative of greater problem with tinnitus.

SECONDARY OUTCOMES:
The Tinnitus Questionnaire (Chinese version) (TQ-CH) scores | Change from baseline value at 3 months, 6 months and 12 months after the first day of treatment will be measured.
  The TQ-CH is a 52-item questionnaire which assesses five dimensions of tinnitus complaint: emotional distress; auditory perceptual difficulties; intrusiveness; sleep disturbance; and somatic complaints. The total TQ score ranges 0 - 104, the higher score is indicative of greater problem with tinnitus.
The Tinnitus Handicap Inventory (Chinese version) (THI-CH) scores | Change from baseline value at 3 months, 6 months and 12 months after the first day of treatment will be measured.
  The THI-CH is a reliable 25-item self-administered Chinese QoL tool that quantifies the impact of tinnitus on daily living. The total THI score ranges 0 - 100, the higher score is indicative of greater tinnitus handicap.
Self-rated Visual Analogue Scale (VAS) on tinnitus loudness | Change from baseline value at 3 months, 6 months and 12 months after the first day of treatment will be measured.
  The subjects will be asked to rate the perceived loudness of their tinnitus on VAS, with "inaudible" (scale rating value = 0) and "very loud" (scale rating value = 100) as reference points for the ends of the scale. The higher rating is indicative of louder tinnitus.
Tinnitus loudness matches at the tinnitus frequency and at 1000 Hz | Change from baseline values at 3 months, 6 months and 12 months after the first day of treatment will be measured.
  Tinnitus loudness matches will be done according to Vernon and Meikle's procedure
The Chinese Hospital Anxiety and Depression Scale (HADS) | Change from baseline value at 3 months, 6 months and 12 months after the first day of treatment will be measured.
  The Chinese HADS is a 14-item questionnaire that consists of two subscales that measure anxiety and depression. It serves as an outcome measure targeting psychological and mental health effects.

CONTACTS AND LOCATIONS:
Overall Officials: Anna CS KAM, AuD, Principal Investigator — The Education University of Hong Kong
Locations (1):
- The Education University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kam ACS. Efficacy of Amplification for Tinnitus Relief in People With Mild Hearing Loss. J Speech Lang Hear Res. 2024 Feb 12;67(2):606-617. doi: 10.1044/2023_JSLHR-23-00031. Epub 2024 Jan 25. PMID 38271299